CLINICAL TRIAL: NCT05434858
Title: Imagery as Biomarker of Imminent Transition From Asymptomatic Hyper Uricemia to Gout
Brief Title: Imagery as Biomarker of Gout
Acronym: TIGER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Collaborators: Auckland University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC-P0097
Record Dates: First submitted 2022-06-14; First posted 2022-06-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hyperuricemia
Keywords: Dual-energy computed tomography; hyperuricemia; gout; monosodium urate crystals
MeSH Terms: conditions — Hyperuricemia; Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient at high risk for gout due to elevated serum urate concentrations (≥ 8 mg/dL) (Experimental): Patients at high risk for gout due to elevated serum urate concentrations (≥ 8 mg/dL) will be included.
  The participants included will be followed for a period of 60 months, with an initial visit, a final visit as well as an additional visit in case of suspicion of gout.
  The presence of symptoms suggestive of gout will be evaluated during regular contact with the participants: a telephone call every 6 months as well as a postal or electronic mail every 3 months. Participants will be asked to contact the investigator if new symptoms or relevant medical events occur.
  Blood (32.5 ml maximum) and urine (4 ml) samples will be taken from participants who have given their specific consent for a biological collection with a particular genetic aim.
  Interventions: Other: Dual-energy CT (DECT) and ultrasound

INTERVENTIONS:
Other: Dual-energy CT (DECT) and ultrasound — DECT and ultrasound will be performed to clarify the pathological mechanisms responsible for the transition from asymptomatic crystalline deposition to gout, and the mechanisms involved in the transition from hyperuricemia to de novo crystalline deposition.

SUMMARY:
The objective of this study is to determine whether MSU crystal deposits visualized on ultrasound and/or DECT are associated with the development of symptomatic gout (according to ACR 2015 / EULAR criteria) over 5 years in hyperuricemic individuals.

DETAILED DESCRIPTION:
Cross-sectional studies have shown that 17% to 86% of people with apparently asymptomatic hyperuricemia have ultrasound evidence of monosodium urate (MSU) crystal deposition. These observations suggest that this deposition constitutes the first stage of the clinical gout syndrome, which has led to a revised model of disease progression and staging. However, no longitudinal studies have been undertaken to determine whether such findings are needed for the development of gout, or to investigate pathological mechanisms responsible for the transition from asymptomatic crystalline deposit to gout. Only a prospective cohort study of people at risk who are carefully and regularly followed can answer such questions.

Dual-energy computed tomography (DECT) and ultrasound are the two imaging techniques that allow the visualization and quantification of MSU crystals. Ultrasound is the most widely used technique; it allows the identification of the deposit of crystals of on the surface of the cartilage (double contour sign) and of the tophi. The DECT can detect the deposition of MSU crystals in soft tissues as long as the amount of crystals exceeds the spatial resolution of the machine (about 250 μm).

The international collaborative study TIGER (Transitions in gout research study) aims to address the question of the predictive value of the deposition of MSU crystals "silent" in the development of gout, through an international cohort (7 countries) including 907 asymptomatic hyperuricaemic individuals. These individuals will have initial ultrasounds to investigate the presence of MSU crystal deposits and a 5-year follow-up. Given the aforementioned ultrasound reproducibility issues, DECT analyzes will be added to the baseline assessment of TIGER participants to provide exploratory data on DECT as a potential biomarker for the impending development of gout.

ELIGIBILITY:
Inclusion Criteria:

* Serum urate level ≥ 80 mg/L on inclusion,
* No current or previous clinical symptoms of gout (including clinically apparent flares or tophus),
* Between 18 and 80 years old,
* Able to give informed consent.

Exclusion Criteria:

* GFR (glomerular filtration rate) <30 ml / min / 1.73 m² or dialysis,
* Serious illness with a poor prognosis of less than 5 years,
* Autoimmune inflammatory arthritis,
* Change of geographical area within 5 years,
* Previous analysis of synovial fluid showing crystals of MSU,
* Presence of subcutaneous tophi,
* Taking a hypouricaemic treatment (allopurinol, probenecid, benzbromarone, febuxostat, lesinurad), canakinumab, anakinra or colchicine,
* Uricemia observed only after an acute decompensation of comorbidity
* Pregnant or breastfeeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2029-09-09 (Estimated)

PRIMARY OUTCOMES:
Odd ratios and its 95% confidence interval for the development of gout | 60 months
  Development of symptomatic gout will be determined according to ACR/EULAR 2015 criteria at any time during the follow-up period. This scale is based on clinical, laboratory and imaging parameters. More than 8 points is considered as Gout. 0 is considered as absence of gout

SECONDARY OUTCOMES:
Time until development of gout symptoms | 60 months
  Time from initial visit to onset of symptomatic gout
Odd Ratio and its 95% confidence interval for gout development according to MSU volume | 60 months
Odd Ratio and its 95% confidence interval for comorbidities development according to MSU volume | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Pascart, MD, PhD, Principal Investigator — Lille Catholic University
Locations (1):
- Lille Catholic Hospital, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No